CLINICAL TRIAL: NCT01592279
Title: GLP-1 Analogue Treatment in Uncontrolled Type 1 Diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 597-11
Record Dates: First submitted 2012-04-30; First posted 2012-05-07 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-04

CONDITIONS: Uncontrolled Type 1 Diabetic Patients
MeSH Terms: interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- liraglutide (Experimental)
  Interventions: Drug: liraglutide
- Insulin injections (Active Comparator)
  Interventions: Drug: Insulin injections

INTERVENTIONS:
Drug: liraglutide
  Arms: liraglutide
Drug: Insulin injections
  Arms: Insulin injections

SUMMARY:
The new incretin-based therapies offer appealing advantages over existing drugs. Aside from glucose dependent insulin secretion and a proven glucose lowering efficacy, they have other concomitant beneficial effects, such as low risk of hypoglycemia, inhibition of the glucagon secretion with maintenance of counter-regulatory mechanism, promotion of weight loss, and possible cardiovascular benefits (improvement of lipid profile, blood pressure, endothelial and myocardial function). The glucose lowering effects resulting from the inhibition of glucagon secretion and the gastric emptying rate could be of clinical importance in type 1 diabetes.

The rationale behind the use of GLP-1 analogues in the treatment of type 1 diabetes relies on the assumption that these drugs, in addition to their action on insulin secretion and glucose regulation, may be effective in preserving and even expanding the β-cell mass. This class of drugs may represent an entirely new approach to the treatment of type 1 diabetes, focused on protection and preservation of β-cells. These therapies have the opportunity to interfere with the disease progression if used as an early intervention, when enough β-cell mass/ function can still be preserved or restored.

Hypothesis:

GLP-1 analogue (liraglutide) will improve glycemic control as measured by HbA1c in uncontrolled type 1 diabetic patients. The investigators expect a reduction of 1% in HbA1C from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. HbA1C ≥ 8 at screening and at qualification
2. Not treated with GLP-1 analogue

Exclusion Criteria:

1. Moderate and sever hypoglycemia
2. Creatinin > 2
3. amylase or lipase > 3xULN
4. Calcitonin > 10 pg/ml or Stimulated Calcitonin > 50 pg/ml in women or 80 pg/ml in men
5. ALT or AST > 3X ULN

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The primary end point is the change in HbA1C relative to baseline after 3 months treatment with liraglutide in uncontrolled type 1 diabetic patients. The expected change is 1% reduction from baseline. | the change in HbA1C relative to baseline after 3 months treatment with liraglutide in uncontrolled type 1 diabetic patients.

SECONDARY OUTCOMES:
Endogenous insulin secretion and residual β-cell function estimated by the value of C-peptide | the change in C-peptide relative to baseline after 3 months treatment with liraglutide in uncontrolled type 1 diabetic patients